CLINICAL TRIAL: NCT01596842
Title: Effect of Omega-3 Fatty Acid on Vitamin D Activation in Hemodialysis Patients
Brief Title: Effect of Omega-3 Fatty Acid on Vitamin D Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, WON SUK AN, Principal Investigator, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAU-12-073
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hemodialysis Patients; Vitamin D Insufficiency; Vitamin D Deficiency
Keywords: Omega-3 fatty acid; vitamin D; ergocalciferol; hemodialysis
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Omacor; Olive Oil; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acid (Active Comparator)
  Interventions: Drug: Omega-3 fatty acid ethylester 90; Other: cholecalciferol
- Olive oil (Placebo Comparator)
  Interventions: Other: Olive oil; Other: cholecalciferol

INTERVENTIONS:
Drug: Omega-3 fatty acid ethylester 90 — Omega-3 fatty acid ethylester 90, Dosage form :1g soft capsule, Dosage : one capsule, thrice a day, Duration : 12 weeks
  Other Names: Omacor®
  Arms: Omega-3 fatty acid
Other: Olive oil — Olive oil, Dosage form :1g soft capsule, Dosage : one capsule, thrice a day, Duration : 12 weeks
  Arms: Olive oil
Other: cholecalciferol — if baseline 25-hydroxyvitamin D levels are < 15 ng/mL : 10,000IU/week, if baseline 25-hydroxyvitamin D levels are 16-30 ng/mL : 50,000IU/week, Duration : 12 weeks

SUMMARY:
Extra-renal sources of 1, 25-dihydroxyvitamin D can be increased to normal serum 1, 25-dihydroxyvitamin D levels in chronic kidney disease patients after administration of high dose 25-hydroxyvitamin D. The investigators observed that 1, 25-dihydroxyvitamin D concentrations were significantly increased after 3 months of omega-3 FA supplementation compared to baseline levels without 25-hydroxyvitamin D administration in dialysis patients. In this study, the investigators hypothesized that omega-3 FA and 25-hydroxyvitamin D supplementations may increase 1, 25-dihydroxyvitamin D concentrations much more compared to 25-hydroxyvitamin D supplementation only in hemodialysis patients with insufficient or deficient 25-hydroxyvitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated with hemodialysis for at least 6 months with 25-hydroxyvitamin D < 30 ng/mL

Exclusion Criteria:

* Patients with a history of active infection within 3 months,
* Patients with fish oil or omega-3 fatty acid supplementation within 3 months,
* Patients with a history of fish, gelatin, and/or omega-3 fatty acid allergies,
* Patients with a history of hospital admission within 3 months,
* Patients with a history of bleeding within 3 months,
* Patients with thrombocytopenia,
* Patients with current use of warfarin,
* Patients with an albumin level < 3.0 g/dL,
* Patients with malignancy and/or liver cirrhosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Won Suk An, Busan, South Korea

REFERENCES:
- [Derived] Lee SM, Son YK, Kim SE, An WS. The effects of omega-3 fatty acid on vitamin D activation in hemodialysis patients: a pilot study. Mar Drugs. 2015 Jan 28;13(2):741-55. doi: 10.3390/md13020741. PMID 25636157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid | Olive Oil
Started | 10 | 7
Completed | 8 | 7
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Hemodialysis patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acid | Olive Oil | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.3) | 64.4 (8.5) | 62.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: 25-hydroxyvitamin D Levels at 12 Weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Omega-3 Fatty Acid | Olive Oil
Number analyzed (Participants) | 8 | 7
ng/ml | 44.4 (10.8) | 48.9 (5.8)

2. Secondary Outcome: Hemoglobin Levels at 12 Weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Omega-3 Fatty Acid | Olive Oil
Number analyzed (Participants) | 8 | 7
g/dL | 10.3 (0.7) | 11 (1.1)

3. Secondary Outcome: Changes of Calcium Levels
Time Frame: 4 weeks, 8 weeks and 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change of Intact Parathyroid Hormone
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change of Fetuin-A Levels
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change of FGF-23 Levels
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Changes of Phosphorous Levels
Time Frame: 4 weeks, 8 weeks and 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Changes of Erythropoietin Doses
Time Frame: 4 weeks, 8 weeks and 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Changes of Phosphate Binder Doses
Time Frame: 4 weeks, 8 weeks and 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Omega-3 Fatty Acid | Olive Oil
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid (N=10) | Olive Oil (N=7)
vaginal spotting (Reproductive system and breast disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes